CLINICAL TRIAL: NCT03392740
Title: Prophylactic Lisinopril to Prevent Anthracycline Induced Left Ventricular Systolic Dysfunction (PLAID) Study.
Brief Title: Prophylactic Lisinopril to Prevent Anthracycline Cardiomyopathy.
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: PI Andrew Hinojos Left Institution (Genesys) prior to Ascension Acquiring record
Sponsor: Ascension Health (Industry)
Responsible Party: Principal Investigator, Jackie Kirchen, Cardiology Fellow, Ascension Health
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: GHIGHCI2018
Record Dates: First submitted 2018-01-02; First posted 2018-01-08 (Actual); Last update posted 2024-05-20 (Actual); Status verified 2024-05

CONDITIONS: Cardiomyopathy Due to Drug; Heart Failure, Systolic
MeSH Terms: conditions — Heart Failure, Systolic | interventions — Lisinopril

STUDY DESIGN:
Intervention Model Description: Prospective, 1:1 randomized, double-blinded and placebo-controlled clinical trial we plan to enroll patients who are to be treated with anthracycline chemotherapy to either lisinopril or placebo group.
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Lisinopril treatment (Experimental): These patients will be initiated at 5mg lisinopril daily by the research nurse at the time of enrollment. The drug will then be titrated up by the research nurse in a stepwise fashion from 5mg, to 10mg, and then to 20mg once a day every 1 to 3 weeks according to their regular/scheduled next office visits. Blood pressure will be monitored at every visit by the research nurse if it is less than or equal to 90 mmHg
  Interventions: Drug: Lisinopril
- Placebo Oral Tablet (Placebo Comparator): These patients will be started on the placebo medication at the time of enrollment. According to their regular scheduled visits every 1 to 3 weeks, they will meet with the research nurse and be given a new placebo medication to take once a day.
  Interventions: Drug: Placebo Oral Tablet

INTERVENTIONS:
Drug: Lisinopril — Patients will be given lisinopril once a day prior to starting an anthracycline chemotherapy regimen and titrated up in a stepwise fashion, as allowed by patients blood pressure, to a target dose of 20mg daily.
  Arms: Lisinopril treatment
Drug: Placebo Oral Tablet — Patients will be given a look-alike placebo medication once a day prior to starting an anthracycline chemotherapy regimen. They will be given a new placebo medication in a step-wise fashion over period of 1 to 3 weeks.
  Arms: Placebo Oral Tablet

SUMMARY:
The intent of the study is to show the potential benefits of angiotensin converting enzyme inhibitors in preventing anthracycline induced cardiotoxicity.

This is a prospective, randomized, blinded and placebo-controlled clinical trial that will enroll patients who are to be treated with anthracycline chemotherapy (doxorubicin, epirubicin, idrarubicin, or mitoxantone) to either lisinopril or placebo group. The study will be performed at the Genesys Hurley Cancer Institute. The treating oncologist who intends to start the patient on anthracycline chemotherapeutic agent will provide the patient with a recruitment flyer and informed consent form and then referred to the research nurse. Subjects interested in participation, that do not meet any of the exclusion criteria, will be consented and enrolled by the research nurse prior to their first treatment with chemotherapy. Over a period of 1 to 3 weeks the study medication will be titrated in a stepwise fashion to a target of 20 mg daily, maintaining a systolic blood pressure greater than 90 mmHg. A baseline echocardiogram with strain and strain rate imaging will be obtained prior to initiation of anthracycline chemotherapy. Subsequent echocardiograms with strain and strain rate imaging will be performed every 3 months for a total of 12 months.

Patients will be followed for a total of 12 months, starting on the day of enrollment. We intend to recruit a total of 200 patients.

The primary endpoint of this study is a change in change in strain and strain rate parameters prior to, during, and after anthracycline chemotherapy compared to placebo.

Study data will be collected and managed using the Ascension installation of REDCap (Research Electronic Data Capture). REDCap is a secure, web application designed to support data capture for research studies, providing user-friendly web-based case report forms, real-time data entry validation (e.g. for data types and range checks), audit trails and a de-identified data export mechanism to common statistical packages.

Echocardiographic data will be stored in cine-loop format on a private, password protected echocardiogram viewing software and analyzed by a separate blinded cardiologist.

Patients will be evaluated according to the standard oncologic evaluation. The treating oncologist will make decisions on their treatment based on their personal standards and clinical judgement.

DETAILED DESCRIPTION:
To date anthracycline chemotherapy regimens still play a major role in many cancer treatments, approximately 32% of breast cancer patients, 57-70% of elderly lymphoma patients, and 50-60% of childhood cancers survivors are treated with an anthracycline regimen.

Of these patients, approximately 9-24%% of patients on anthracycline chemotherapy will develop anthracycline cardiomyopathy and the majority will present with signs and/or symptoms within the first 12 months of starting chemotherapy. The onset of anthracycline cardiomyopathy, even asymptomatic, not only negatively impacts the cardiac outcome of cancer patients, but also limits their therapeutic opportunities to less aggressive and, consequently, less effective therapies

There is limited evidence based research for treatment of anthracycline induced cardiomyopathy and is mainly targeted towards standard heart failure therapy. In 2006, Cardinale et al. found early treatment of myocardial cell injury, as defined by a rise in troponin, with enalapril prevents left ventricular ejection fraction decrease as well as the occurrence of cardiac events. Subsequently in 2010, Cardinale et al. also found that treatment of anthracycline cardiomyopathy with standard heart failure therapy (enalapril, carvedilol) at the onset of cardiomyopathy, defined as ejection fraction of ≤ 45%, lead to complete recovery of left ventricular ejection fraction and improved cardiac outcomes. Indeed, much of the research has been focused on management of patients who develop early signs of left ventricular dysfunction. Unfortunately, despite this strategy up to 11% still go on to develop New York Heart Association class 3 or 4 heart failure symptoms.

A crucial issue remains is whether or not, and eventually how, to treat patients still asymptomatic who do not yet demonstrate left ventricular dysfunction. Lisinopril use has been well studied in patients with systolic heart failure and is a class I indication in all patients with an ejection fraction of <40 %. Randomized control trials have established their benefit in reducing morbidity and mortality in heart failure with reduced ejection fraction. Since anthracycline induced-cardiotoxicity has a significant impact on overall prognosis in cancer patients and despite treatment after the development of left ventricular dysfunction from anthracyclines will still result in a large amount of the patient population developing heart failure, there is an urgent need in prophylactic treatment in preventing anthracycline-induced left ventricular dysfunction.

Thus, the intent of our study is to show the potential benefits of angiotensin converting enzyme inhibitors in preventing anthracycline induced cardiotoxicity.

This is a prospective, randomized, blinded and placebo-controlled clinical trial that will enroll patients who are to be treated with anthracycline chemotherapy (doxorubicin, epirubicin, idrarubicin, or mitoxantone) to either lisinopril or placebo group. The study will be performed at the Genesys Hurley Cancer Institute. The treating oncologist who intends to start the patient on anthracycline chemotherapeutic agent will provide the patient with a recruitment flyer and informed consent form and referred to the research nurse. Subjects interested in participation, that do not meet any of the exclusion criteria, will be consented and enrolled by the research nurse prior to their first treatment.

The study protocol is outlined below.

Enrollment (Performed by the Genesys Hurley Cancer Institute research nurse):

* Baseline characteristics will be obtained including: age, comorbidities, medications, family history of cardiovascular disease, smoking status, and body measurements (height and weight).
* Patient will be sent for echocardiogram to be performed at Genesys Heart Institute
* Patient will be randomized to either study or placebo drug. If in the study group, they will be started on lisinopril 5mg oral tablet once a day. If in the placebo group, they will be started on the placebo drug by the research pharmacy

First day of treatment (typically 1-3 weeks after enrollment). The following will be performed by the Genesys Hurley Cancer Institute research nurse and research pharmacist:

* Vital signs will be taken and recorded
* Subject will be screened for any side effects from study drug. If side effects are noted the Genesys Hurley Cancer Institute research nurse will contact the study investigator (Andrew Hinojos) for further instruction.
* If the subjects systolic blood pressure is above 90 mmHg, they will be instructed to take 2 tablets of lisinopril 5mg once a day (equivalent to 10mg once a day) or instructed to take 2 tablets of placebo drug once a day to maintain the blind.
* If the subjects systolic blood pressure is below 90 mmHg, they will be taken off the study drug (Lisinopril or placebo) and removed from the study. The study investigator will be contacted to evaluate for adverse events

Follow up visit (Typically 1-3 weeks after first treatment). The following will be performed by the Genesys Hurley Cancer Institute research nurse and research pharmacist:

* Vital signs will be taken and recorded
* Subject will be screened for any side effects from study drug. If side effects are noted the research nurse will contact the study investigator (Andrew Hinojos) for further instruction
* If the subjects systolic blood pressure is above 90 mmHg and they are currently taking 2 tablets of lisinopril 5mg once a day (equivalent to 10mg once a day), they will be instructed to take 4 tablets of lisinopril 5mg once a day (equivalent to 20mg once a day). The placebo group will be instructed to take 4 tablets of placebo drug once a day to maintain blind.
* If the subjects systolic blood pressure is below 90 mmHg and they are currently taking 2 tablets of lisinopril 5mg once a day (equivalent to 10mg once a day), they will instructed to decrease to 1 tablet lisinopril 5mg once a day. They will be maintained on that dose of lisinopril 5mg once a day for 12 months. Those in the placebo group, the study investigator will be contacted to rule out adverse events. If no adverse events, they will be instructed to take 1 tablet of placebo drug once a day.

Second treatment (Typically 1-3 weeks after first treatment). The following will be performed by the Genesys Hurley Cancer Institute research nurse and research pharmacist:

* Vital signs will be taken and recorded
* Subject will be screened for any side effects from study drug. If side effects are noted the research nurse will contact the study investigator (Andrew Hinojos) for further instruction.
* If the subjects systolic blood pressure is above 90 mmHg and they are taking 4 tablets of lisinopril 5mg once a day (equivalent to 20mg once a day). They will be maintained at this dose for 12 months.
* If the subjects systolic blood pressure is less than or equal to 90 mmHg and they are currently taking 4 tablets of lisinopril 5mg once a day, they will be instructed to take 2 tablets of lisinopril 5mg once a day (equivalent to 10mg once a day). They will be maintained on this regimen for 12 months
* If the subject is in the placebo group and the systolic blood pressure is less than or equal to 90 mmHg: The study investigator will be contacted to rule out adverse events. If no adverse events, they will be instructed to take 2 tablet of placebo drug once a day
* If the subject is on 1 tablet of lisinopril 5mg once a day: If systolic blood pressure is above 90 mmHg they will be maintained at this dose for 12 months. If systolic blood pressure is 90mmHg or below they will be taken off the study drug and remove from the study

Echocardiograms with strain and strain rate will be performed at enrollment, 3 months, 6 months, 9 months, and 12 months intervals from enrollment date.

The Genesys Hurley Cancer Institute Research Pharmacy will be responsible for administration of the placebo and the study drug. They will be aware ("unblinded") of the patients participation in either the study or placebo group. They will be responsible for maintaining that the investigators and research team remain "blind" to the patients allocated group by administration of the placebo, which is formulated to appear similar to the study drug(s).

The research nurse, oncology team, cardiology team, and study investigators will be unaware of which drug the subject is receiving which will be made confidential with the help of the GHCI research pharmacy and our database management system, RedCap.

If any potential drug interactions are identified or the patients blood pressure is persistently low, which cannot be resolved by the blinded principal investigator, we have designated an "unblinded" research investigator, Victor Medina to resolve these issues.

The primary endpoint of this study is a change in change in strain and strain rate parameters prior to, during, and after anthracycline chemotherapy compared to placebo.

Secondary outcomes are based on the American Society of Echocardiography consensus on cancer therapeutics-related cardiac dysfunction (CTRCD). CTRCD is defined as a decrease in ejection >10% below 53% with at least 2 signs and symptoms of heart failure (lower extremity swelling, elevated jugular venous pulsation, orthopnea, paroxysmal nocturnal dyspnea, dyspnea on exertion). Those with a baseline ejection fraction <53% at baseline will be placed in the secondary endpoint if their ejection fraction decreases by >10% from their baseline with at least 2 signs and/or symptoms of heart failure. We will also examine, subclinical anthracycline cardiomyopathy defined as a decrease in ejection fraction >10% below 53% without signs and/or symptoms of heart failure. In those with a baseline ejection fraction <53% at baseline will be placed in the secondary endpoint if their ejection fraction decreases by >10% from their baseline without at least 2 signs and/or symptoms of heart failure. We will also examine the occurrence of cardiac events during the 1-year follow-up defined as death from any cause, death resulting from a cardiac cause, acute pulmonary edema, overt heart failure, and life-threatening arrhythmias requiring treatment.

Based on a predetermined estimation that the treatment decreases the event rate by 50% (10% versus 20%), the study investigators intend to recruit approximately 95 patients per group.

Blind conventional 2 dimensional echocardiography will be performed using standard commercially available equipment. Imaging will be conducted with patients either supine or in the left lateral decubitus position. Data will be acquired using a 3.5-MHz transducer in the apical (2- and 4-chamber and apical long axis) and parasternal (long and short axis) views according to the American Society of Echocardiography. Transmitral flow velocity signals will be obtained in the four-chamber view by placing a 2-mm pulsed doppler sample volume at the tips of the valve leaflets, aligned with the left ventricular inflow by color flow imaging. Peak early (E) and late diastolic (A) velocities, E-wave deceleration time, ratio of E and A wave and A-wave duration will be measured.

A comprehensive assessment of the strain and strain rate for the left ventricular myocardium using tissue Doppler-based imaging (TDI). Standard 2D gray-scale images of the left ventricle with a mean frame rate of 90 ± 5 frames per second at conventional apical 2- and 4-chamber views will be acquired. The parameters measured will be the peak systolic velocity, early and late systolic velocities, early and late diastolic velocities. Basal values are considered to represent the best reproducibility for TDI-based strain assessment. Peak systolic longitudinal strain and strain-rate parameters will be calculated and derived from four segments of the two apical chambers (2- and 4-chamber views).

Study data will be collected and managed using the Ascension installation of REDCap (Research Electronic Data Capture). REDCap is a secure, web application designed to support data capture for research studies, providing user-friendly web-based case report forms, real-time data entry validation (e.g. for data types and range checks), audit trails and a de-identified data export mechanism to common statistical packages.

Echocardiographic data will be stored in cine-loop format on a private, password protected echocardiogram viewing software and analyzed by a separate blinded cardiologist.

Patients will be evaluated according to the standard oncologic evaluation. The treating oncologist will make decisions on their treatment based on their personal standards and clinical judgement.

Patients who develop anthracycline induced heart failure will be treated according to the treating oncologist and clinical scenario.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with a type of cancer and intended to be on an anthracycline chemotherapy regimen by treating oncologist.

Exclusion Criteria:

* Inability or unwillingness to give informed consent
* Subjects with a contraindication to angiotensin converting enzyme inhibitors such as history of angioedema or hypersensitivity related to previous treatment with an angiotensin converting enzyme inhibitor
* Subjects with a history of hereditary or idiopathic angioedema
* Subjects currently taking aliskiren (major drug interaction-)
* Subjects currently taking a neprilysin inhibitor (e.g. sacubitril or entresto)
* Subjects already on treatment with angiotensin converting enzyme inhibitors, or taking lithium
* Renal insufficiency defined as creatinine clearance <30
* Women <50 who capable of child bearing who have not had surgical contraception such as hysterectomy or tubal ligation
* Oncologic life expectancy shorter than 12 months
* Systolic blood pressure <90 mmHg prior to enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-03-15 (Estimated); Primary Completion 2018-12-15 (Actual); Study Completion 2018-12-15 (Actual)

PRIMARY OUTCOMES:
Change in strain rate from baseline | 12 months from enrollment
  The primary outcome is a change in strain and strain rate from baseline echocardiogram

SECONDARY OUTCOMES:
Heart failure and left ventricular dysfunction | 12 months from enrollment
  A decrease in ejection fraction >10% below 53% from baseline with at least 2 signs and symptoms of heart failure (lower extremity swelling, elevated jugular venous pulsation, orthopnea, paroxysmal nocturnal dyspnea, dyspnea on exertion). In those with an ejection fraction <53% at baseline will be placed in the primary endpoint if their ejection fraction decreases by >10% from their baseline with at least 2 signs and/or symptoms of heart failure.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Hinojos, DO, Principal Investigator — Genesys Regional Medical Center Department of Education
Locations (1):
- Genesys Regional Medical Center, Grand Blanc, Michigan, United States

IPD SHARING:
Plan to Share IPD: Undecided
It is undecided at this point and there currently is not a plan to make individual participant data (IPD) collected in this study available to other researchers.

REFERENCES:
- [Background] McGowan JV, Chung R, Maulik A, Piotrowska I, Walker JM, Yellon DM. Anthracycline Chemotherapy and Cardiotoxicity. Cardiovasc Drugs Ther. 2017 Feb;31(1):63-75. doi: 10.1007/s10557-016-6711-0. PMID 28185035
- [Background] Bird BR, Swain SM. Cardiac toxicity in breast cancer survivors: review of potential cardiac problems. Clin Cancer Res. 2008 Jan 1;14(1):14-24. doi: 10.1158/1078-0432.CCR-07-1033. PMID 18172247
- [Background] Cardinale D, Colombo A, Lamantia G, Colombo N, Civelli M, De Giacomi G, Rubino M, Veglia F, Fiorentini C, Cipolla CM. Anthracycline-induced cardiomyopathy: clinical relevance and response to pharmacologic therapy. J Am Coll Cardiol. 2010 Jan 19;55(3):213-20. doi: 10.1016/j.jacc.2009.03.095. PMID 20117401
- [Background] Yeh ET, Tong AT, Lenihan DJ, Yusuf SW, Swafford J, Champion C, Durand JB, Gibbs H, Zafarmand AA, Ewer MS. Cardiovascular complications of cancer therapy: diagnosis, pathogenesis, and management. Circulation. 2004 Jun 29;109(25):3122-31. doi: 10.1161/01.CIR.0000133187.74800.B9. PMID 15226229
- [Background] Seicean S, Seicean A, Plana JC, Budd GT, Marwick TH. Effect of statin therapy on the risk for incident heart failure in patients with breast cancer receiving anthracycline chemotherapy: an observational clinical cohort study. J Am Coll Cardiol. 2012 Dec 11;60(23):2384-90. doi: 10.1016/j.jacc.2012.07.067. Epub 2012 Nov 7. PMID 23141499
- [Background] Gulati G, Heck SL, Ree AH, Hoffmann P, Schulz-Menger J, Fagerland MW, Gravdehaug B, von Knobelsdorff-Brenkenhoff F, Bratland A, Storas TH, Hagve TA, Rosjo H, Steine K, Geisler J, Omland T. Prevention of cardiac dysfunction during adjuvant breast cancer therapy (PRADA): a 2 x 2 factorial, randomized, placebo-controlled, double-blind clinical trial of candesartan and metoprolol. Eur Heart J. 2016 Jun 1;37(21):1671-80. doi: 10.1093/eurheartj/ehw022. Epub 2016 Feb 21. PMID 26903532
- [Background] Packer M, Poole-Wilson PA, Armstrong PW, Cleland JG, Horowitz JD, Massie BM, Ryden L, Thygesen K, Uretsky BF. Comparative effects of low and high doses of the angiotensin-converting enzyme inhibitor, lisinopril, on morbidity and mortality in chronic heart failure. ATLAS Study Group. Circulation. 1999 Dec 7;100(23):2312-8. doi: 10.1161/01.cir.100.23.2312. PMID 10587334
- [Background] Yancy CW, Jessup M, Bozkurt B, Butler J, Casey DE Jr, Colvin MM, Drazner MH, Filippatos GS, Fonarow GC, Givertz MM, Hollenberg SM, Lindenfeld J, Masoudi FA, McBride PE, Peterson PN, Stevenson LW, Westlake C. 2017 ACC/AHA/HFSA Focused Update of the 2013 ACCF/AHA Guideline for the Management of Heart Failure: A Report of the American College of Cardiology/American Heart Association Task Force on Clinical Practice Guidelines and the Heart Failure Society of America. J Am Coll Cardiol. 2017 Aug 8;70(6):776-803. doi: 10.1016/j.jacc.2017.04.025. Epub 2017 Apr 28. No abstract available. PMID 28461007
- [Background] Geisberg CA, Sawyer DB. Mechanisms of anthracycline cardiotoxicity and strategies to decrease cardiac damage. Curr Hypertens Rep. 2010 Dec;12(6):404-10. doi: 10.1007/s11906-010-0146-y. PMID 20842465
- [Background] Georgakopoulos P, Roussou P, Matsakas E, Karavidas A, Anagnostopoulos N, Marinakis T, Galanopoulos A, Georgiakodis F, Zimeras S, Kyriakidis M, Ahimastos A. Cardioprotective effect of metoprolol and enalapril in doxorubicin-treated lymphoma patients: a prospective, parallel-group, randomized, controlled study with 36-month follow-up. Am J Hematol. 2010 Nov;85(11):894-6. doi: 10.1002/ajh.21840. PMID 20872550